CLINICAL TRIAL: NCT05677594
Title: Multi-parametric Biomarker Development to Predict Malignant Conversion in Patients With Neurofibromatosis Type 1
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Neurofibromatosis Therapeutic Acceleration Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00268132
Record Dates: First submitted 2022-12-09; First posted 2023-01-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis 1; Malignant Peripheral Nerve Sheath Tumor (MPNST) of Soft Tissue (Diagnosis); Atypical Neurofibroma
Keywords: Whole Body Magnetic Resonance Imaging; Biomarker
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibrosarcoma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Whole Body Magnetic Resonance Imaging — Magnetic resonance imaging of the entire body from skull base through distal thighs/knees without contrast material

SUMMARY:
The goal of this prospective observational study is to learn about the utility of imaging and clinical features in patients with Neurofibromatosis type 1 categorized as high risk for the development of malignant peripheral nerve sheath tumors.

The main objectives are:

* To evaluate the prevalence, multi-parametric imaging features of distinct nodular lesions ("DNLs") and natural history in people with NF1 with clinical and genetic features deemed "high-risk" for malignancy.
* To assess the relationship between individual clinical, genetic and imaging factors that have been suggested to be risk factors for malignant peripheral nerve sheath tumors (MPNST) and the confirmation of atypical neurofibromas (aNF)/ atypical neurofibromatous neoplasm of unknown biologic potential (ANNUBP) or MPNST on pathology.

In this research study, the participants will be asked to undergo whole body MRI, provide blood sample and clinical evaluation annually.

DETAILED DESCRIPTION:
Patients with the autosomal dominant genetic tumor predisposition syndrome neurofibromatosis type 1 (NF1) have an increased risk of developing both benign and malignant neoplasms throughout life. The most common tumors are peripheral nerve sheath tumors (PNSTs) such as plexiform neurofibromas (pNFs). pNFs are multicellular primary tumors of the peripheral nerve that are histologically benign but often cause significant neurologic morbidity due to involvement of critical nerves. However, the greatest fear is the development of malignant peripheral nerve sheath tumors (MPNSTs). MPNST is an aggressive, treatment resistant sarcoma with a 5-year survival rate of only 15-50% and is the leading cause of death in NF1 patients, especially in those under 50 years of age. An estimated 50% of NF1 patients develop pNFs and the lifetime risk of developing MPNST is 8-13%. The only possible cure for MPNST is complete resection with wide negative margins. This is only feasible if the lesion can be clearly defined and removed without life-threatening morbidity. A major challenge to clearly differentiating between MPNSTs and pNFs is that the vast majority of MPNSTs arise within pNFs. This intimate association makes it hard to distinguish MPNST clinically, radiologically, and pathologically from surrounding benign tissue, thus leading to delayed diagnosis until after symptoms (such as severe pain and loss of neurologic function) have emerged and the chance for cure is greatly diminished or lost. A great deal of time, resource and worry from patients, the patients loved ones and medical providers is dedicated to detecting MPNSTs early at great expense and unclear benefit.

Existing clinical factors and imaging markers of MPNST do not accurately identify patients at risk of developing either MPNST or the patients precursor tumors. Retrospective studies from various centers have suggested several clinical factors associated with the development of MPNST including: number and volume of internal PNSTs, presence of subcutaneous neurofibromas, younger age, presence of pain, microdeletion of the NF1 gene, family and personal history of MPNST, and presence of atypical neurofibromas (aNF)/ANNUBPs. None of the imaging diagnostic tools studied in NF1 patients have been prospectively assessed to identify aNF/ANNUBP. Natural history studies and clinical trials using MRI have identified nodular target lesions within pre-existing pNFs on standard anatomic MRI as potential precursor lesions to MPNST that may represent aNF/ANNUBP. These lesions have been coined "distinct nodular lesions" (DNLs) and described as greater than 3 cm in largest diameter, well demarcated, distinct from the patients underlying tissue (i.e. the surrounding pNF), and lacking the target sign typical of benign pNFs (defined as a central hypointense region on T2-weighted images). In a recent retrospective review of 76 histologically confirmed aNFs, all aNFs fulfilled the criteria for DNLs on MRI and 50 of 56 aNFs with available 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission testing computed tomography (18F-FDG PET/CT) demonstrated elevated maximum standardized uptake value (SUVmax) (>3.5), supporting the hypothesis that DNLs may be the imaging correlate of pre-malignant tumors.

The investigators hypothesize that NF1 patients with aNF/ANNUBP represent a subset of individuals who have not developed cancer yet but who are at high risk of developing a malignancy, possibly in the short term. the investigators further hypothesize that a subset of DNLs are imaging correlates of aNF/ANNUBP that can be characterized with advanced imaging techniques such as Diffusion weighted imaging (DWI) and 18F-FDG PET/CT. Imaging identification of ANNUBPs and characterization of DNLs will enable early diagnosis and management of lesions destined to become malignant, thereby potentially dramatically improving outcomes for People with NF1 at highest risk for development of MPNST.

Defining the prevalence of DNL in a population clinically to be at high-risk for future development of malignancy, the behavior of DNLs over time and the multi-parametric imaging features of DNLs will allow the generation of imaging markers to: (1) identify the specific lesions at highest risk for malignancy in a sea of lesions, (2) understand the biologic significance of these lesions and, (3) create the data about the optimal imaging marker for these lesions to inform evidence based guidelines for imaging in people with NF1.

2. Objectives (include all primary and secondary objectives):

* To evaluate the prevalence, multi-parametric imaging features of distinct nodular lesions "DNLs" and natural history in people with NF1 with clinical and genetic features deemed "high-risk" for malignancy.
* To assess the relationship between individual clinical, genetic and imaging factors that have been suggested to be risk factors for MPNST and the confirmation of aNF/ANNUBP or MPNST on pathology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are person (age > 6 years) with clinical diagnosis of NF1, ability to undergo whole body MRI without intravenous contrast material considered "high-risk" for MPNST.

The term "high risk" is defined as:

* high pNF burden defined as 1 pNF > 3 cm or > 1 pNF
* diagnosis of whole-gene deletion ("microdeletion") of the NF1 gene on genetic testing
* prior history of atypical or malignant PNST
* family or personal history of MPNST or atypical PNST
* prior radiation treatment

Exclusion Criteria:

* Pregnancy
* inability to tolerate MRI or 18F-FDG-PET/CT imaging without anesthesia
* ongoing NF1-related intervention (including systemic steroids) or therapy that may alter the anatomic, metabolic or functional MRI appearance of the PNSTs.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: High risk persons with NF1 based on genetic testing (microdeletion, family/personal history of atypical NF, ANNUBP, MPNST, prior radiation treatment, large plexiform neurofibroma burden)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of distinct nodular lesions in people with NF1 associated pNF | 4 years
  Prevalence of distinct nodular lesions in people with NF1 associated pNF and clinical or genetic factors that are hypothesized to be "high risk" for MPNST

SECONDARY OUTCOMES:
Imaging features of distinct nodular lesions | 4 years
  The imaging characteristics of DNL over time
Incidence of new distinct nodular lesions | 4 years
  Incidence of new DNLs over time (in both people who do and do not have DNL on initial imaging)
Imaging features of pNF | 4 years
  The imaging characteristics of pNF (independent of DNL) over time in people hypothesized to be "high risk" for MPNST
Histology of distinct nodular lesions | 4 years
  Frequency of biopsy in people with and without DNL.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Ahlawat, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States